CLINICAL TRIAL: NCT06032143
Title: Doulas as Environmental Educators and Partners Study
Acronym: DEEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Tamarra James-Todd, Primary Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB23-0748
Record Dates: First submitted 2023-07-26; First posted 2023-09-11 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Doulas (Experimental): Doulas randomized to the intervention group will engage in a one-hour online course about exposure to phthalates and the relationship with reproductive health.
  Interventions: Behavioral: Online educational phthalate course
- Control Doulas (Sham Comparator): Doulas randomized to the control group will access a worksheet about an alternative environmental exposure and the relationship with reproductive health.
  Interventions: Behavioral: Control environmental education
- Intervention Pregnant Individuals (Experimental): Pregnant individuals working with intervention doulas will be asked to have a conversation with their doulas about environmental chemicals (phthalates).
  Interventions: Behavioral: Phthalate conversation
- Control Pregnant Individuals (Sham Comparator): Pregnant individuals working with control doulas will be asked to have a conversation with their doulas about environmental chemicals (distinct from phthalates).
  Interventions: Behavioral: Environmental exposures conversation

INTERVENTIONS:
Behavioral: Online educational phthalate course — This is an online course focused on phthalates for reproductive health professionals. It consists of videos from patient, scientist, and OBGYN perspectives describing how phthalates relate to reproductive health. There is also an interactive module and worksheet to facilitate conversations about phthalates with pregnant individuals.
  Arms: Intervention Doulas
Behavioral: Control environmental education — Participants in the control group will receive access to environmental exposures other than phthalates.
  Arms: Control Doulas
Behavioral: Phthalate conversation — Participants in the intervention groups will be asked to engage in conversations about phthalates between doulas/pregnant individuals.
  Arms: Intervention Pregnant Individuals
Behavioral: Environmental exposures conversation — Participants in the intervention groups will be asked to engage in conversations about environmental exposures (other than phthalates) between doulas/pregnant individuals.
  Arms: Control Pregnant Individuals

SUMMARY:
The aims of this project are:

Aim 1: Determine the extent to which an environmental health literacy educational intervention designed for doulas improves their environmental health literacy of endocrine disrupting chemicals (EDCs) in personal care products.

Hypothesis 1a. Doulas who participate in an environmental health literacy course will have a higher environmental health literacy score based on quantitative questionnaire evaluation post-course compared to pre-course.

Hypothesis 1b. Doulas who participate in the environmental health literacy course will have a higher environmental health literacy scores post-course compared to doulas who do not take the environmental health literacy course.

Aim 2: Determine the extent to which pregnant people counseled by doulas with training in environmental health literacy have higher environmental health literacy scores and lower usage of personal care products containing EDCs following doula counseling.

Hypothesis 2a. Compared to pregnant people not counseled by doulas on EDCs in personal care products, pregnant individuals counseled by doulas on these EDCs will have improved scores in environmental health literacy.

Hypothesis 2b. Compared to pregnant people not counseled by doulas on EDCs in personal care products, pregnant individuals receiving counseling will use fewer personal care products associated with containing EDCs based on a validated questionnaire.

Aim 3: Determine whether concentrations of EDC biomarkers decreased after the intervention for the intervention group.

Hypothesis 3: Urinary phthalate metabolite concentrations will be lower post-course compared to pre-course for the intervention group.

DETAILED DESCRIPTION:
Compared to other racial/ethnic groups, non-Hispanic black women have significantly higher concentrations of endocrine disrupting chemicals (EDCs) found in personal care products, including phthalates and parabens These EDCs are linked to a variety of adverse reproductive health outcomes that range from early puberty to preterm birth to hot flashes-all conditions that disproportionately impact black women and their long-term health.

Pregnancy is a particularly sensitive window of exposure to EDCs due to normal physiologic changes that alter the body's lipid and glucose metabolism, vasculature, inflammatory, and coagulation responses. Sadly, pregnancy holds some of the most shocking racial/ethnic health disparities, including a 50% increased risk of preterm birth, up to 2-fold increased risk of preeclampsia, and 3-fold increased risk of maternal mortality. Gaps in health care access have been documented as important contributors to these adverse health outcomes, but little research has evaluated the critical gap in environmental health information, particularly information linked to knowledge, awareness, and action related to EDC exposures. In black pregnant people, doulas have increasingly served an important role in filling health care gaps by providing access, advocacy, support, and education at this sensitive window. Yet, doulas often are not equipped to provide key environmental health information around chemical exposures that are higher in black women. If doulas' environmental health literacy of personal care product EDCs linked to adverse pregnancy outcomes was improved, then pregnant people in their care could benefit from reduced exposure to these chemicals and improved pregnancy outcomes. With this, the investigators intend to leverage the supportive advocacy and educational role doulas provide to black pregnant people to improve EDC environmental health literacy by partnering with Black Millennials 4 Flint organization to 1) educate doulas on EDCs; 2) utilize this newly gained knowledge in a clinical setting for doulas to counsel pregnant people on personal care product EDC chemicals; 3) measure environmental health literacy in doulas and the pregnant people they counsel; 4) evaluate urinary phthalate metabolite concentrations before and after the intervention. To conduct this intervention, the investigators will leverage a personal care product EDC module developed by the Harvard Chan's Environmental Reproductive Justice Lab (PI: Dr. Tamarra James-Todd). The investigators will also utilize an environmental health literacy questionnaire, as well as other previously validated quantitative and qualitative data collection tools. The aims of this project are:

Aim 1: Determine the extent to which an environmental health literacy educational intervention designed for doulas improves their environmental health literacy of EDCs in personal care products Hypothesis 1a. Doulas who participate in an environmental health literacy course will have a higher environmental health literacy score based on quantitative questionnaire evaluation post-course compared to pre-course Hypothesis 1b. Doulas who participate in the environmental health literacy course will have a higher environmental health literacy scores post-course compared to doulas who do not take the environmental health literacy course Aim 2: Determine the extent to which pregnant people counseled by doulas with training in environmental health literacy have higher environmental health literacy scores and lower usage of personal care products containing EDCs following doula counseling Hypothesis 2a. Compared to pregnant people not counseled by doulas on EDCs in personal care products, pregnant individuals counseled by doulas on these EDCs will have improved scores in environmental health literacy Hypothesis 2b. Compared to pregnant people not counseled by doulas on EDCs in personal care products, pregnant individuals receiving counseling will use fewer personal care products associated with containing EDCs based on a validated questionnaire Aim 3: Determine whether concentrations of EDC biomarkers decreased after the intervention for the intervention group.

Hypothesis 3: Urinary phthalate metabolite concentrations will be lower post-course compared to pre-course for the intervention group.

ELIGIBILITY:
Inclusion criteria:

* Doulas currently working with pregnant individuals <30 weeks into their pregnancy
* Pregnant individuals working with doulas who are <30 weeks into their pregnancy

Exclusion criteria:

* Doulas not currently working with pregnant individuals <30 weeks into their pregnancy
* Pregnant individuals working with doulas who are beyond 30 weeks into their pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Baseline phthalate environmental health literacy | Up to 2 weeks
  Measure of phthalate reproductive environmental health literacy via validated scale (pre educational intervention), the Phthalate Environmental Reproductive Health Literacy (PERHL) scale. Scores on the PERHL scale range from 6-31, with a higher score indicating higher environmental health literacy.
Change from baseline phthalate environmental health literacy | Up to 4 weeks
  Measure of phthalate reproductive environmental health literacy via validated scale (post educational intervention), the Phthalate Environmental Reproductive Health Literacy (PERHL) scale. Scores on the PERHL scale range from 6-31, with a higher score indicating higher environmental health literacy.
Baseline urinary biomarkers of phthalate exposure | Up to 2 weeks
  Collected via urine samples, measure of previous phthalate exposures for urinary phthalate metabolite concentrations using a standard panel, measuring 16 urinary phthalate metabolites and their replacements (Cyclohexane-1,2-dicarboxylic acid mono carboxyisooctyl ester (CX-MINCH), mono-2-ethyl-5- carboxypentyl terephthalate (MECPTP), mono-2-ethyl-5-hydroxyhexyl terephthalate (MEHHTP), Cyclohexane-1,2-dicarboxylic acid mono hydroxyisononyl ester (OH-MINCH), mono-n-butylphthalate (mBP), mono-benzyl phthalate (mBzP), mono-carboxy isononyl phthalate (mCnP), mono-carboxy octyl phthalate (mCOP), mono (3-carboxypropyl) phthalate(mCPP), mono-(2-ethyl-5-carboxypentyl) phthalate (mECPP), mono (2-ethyl-5-hydroxyhexyl) phthalate (mEHHP), mono ethyl hexyl phthalate (mEHP), mono (2-ethyl-5-oxohexyl) phthalate (mEOHP), monoethyl phthalate (mEP), mono-isononyl phthalate (mNP), mono-isobutyl phthalate (miBP), and assayed using a modified method from the Centers for Disease Control and Prevention.
Change in urinary biomarkers of phthalate exposure | Up to 4 weeks
  Collected via urine samples, measure of previous phthalate exposures. We will evaluate urine samples for urinary phthalate metabolite concentrations using a standard panel, measuring 16 urinary phthalate metabolites and their replacements (CX-MINCH, MECPTP, MEHHTP, OH-MINCH, mBP, mBzP, mCnP, mCOP, mCPP, mECPP, mEHHP, mEHP, mEOHP, mEP, mNP, miBP), and assayed using a modified method from the Centers for Disease Control and Prevention. Briefly, HPLC-MS/MS ESI is conducted based on the CDC's Phthalate Metabolites in Urine Method No: 6306.03. We will also calculate the molar sums of SG-adjusted metabolites representing metabolites related to parent compound DEHP (i.e., ΣDEHP = (mEHP/278) + (mEHHP/294) + (mEOHP/292) + (mECPP/308)) and personal care product (PCP)-associated phthalates (i.e., ΣPCP = (mBP/222) + (miBP/222) + (mEP/194)). Units for all metabolites will be ng/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard T.H. Chan School of Public Health, Boston, Massachusetts, United States